CLINICAL TRIAL: NCT06041139
Title: Visual Outcomes and Patient Satisfaction With Bilateral PanOptix Verses Bilateral Synergy
Status: Completed | Type: Observational
Sponsor: Berkeley Eye Center (Other)
Responsible Party: Sponsor
Other Study IDs: 69881171
Record Dates: First submitted 2022-07-13; First posted 2023-09-18 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pseudophakia
Keywords: Pseudophakia; Alcon PanOptix; Johnson & Johnson Tecnis Synergy
MeSH Terms: conditions — Pseudophakia | interventions — Visual Acuity; Glare

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Alcon PanOptix: Patients will have had bilateral implantation of PanOptix IOLs with the toric and/or non-toric models at the time of uncomplicated cataract surgery.
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Defocus Curve; Diagnostic Test: Halo and Glare testing; Other: Patient Questionnaires
- Johnson & Johnson Synergy: Patients will have had bilateral implantation of Synergy IOLs with the toric and/or non-toric models at the time of uncomplicated cataract surgery.
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Defocus Curve; Diagnostic Test: Halo and Glare testing; Other: Patient Questionnaires

INTERVENTIONS:
Diagnostic Test: Visual Acuity — Measurement of distance, intermediate and near visual acuity.
Diagnostic Test: Defocus Curve — Measurement of visual acuity performed from +1.00 to -4.00 in 0.50 diopter steps and with +0.25 and -0.25 added.
Diagnostic Test: Halo and Glare testing — Measurement to quantify degree of visual loss caused by either halo and/or glare.
  Other Names: VS Halo & Glare (visu-med.com)
Other: Patient Questionnaires — Patients will complete a series of questionnaires to record self-reported visual disturbances, visual acuity satisfaction, level of spectacle independence and any issues with glare, halos, and/or starbursts.
  Other Names: IOLSAT, QUVID and Self-Reported Visual Disturbance Questionnaire

SUMMARY:
Background:

* The Tecnis Synergy intraocular lens (IOL) has a claim to allow patients to experience continuous high-contrast vision from far through near even in low-light conditions.
* A J&J-sponsored post marketing study done outside of the US claim superiority of range of vision for the Tecnis Synergy IOL over the PanOptix IOL.

Hypothesis:

* Patients with bilateral Panoptix IOLs have non-inferior distance, intermediate, and near visual acuity compared to patients with bilateral Synergy IOLs in both photopic and mesopic conditions with less glare, haloes, and/or starbursts.

Unmet Medical Need:

* There is a need to look at patient visual outcomes and the visual disturbance profile comparing trifocal technology with combined EDOF/Bifocal technology in the United States.

DETAILED DESCRIPTION:
* This is a non-interventional single center, two-arm comparative study of the outcomes for patients following successful, uncomplicated cataract surgery.
* There will be 155 subjects enrolled in each arm (310 subjects total).
* Consecutive screening will be used for enrollment beginning from the first bilateral IOL implanted.
* All testing will be at a single site with subjects coming from 4 surgeons (all use similar surgical technique) at that site.
* Each surgeon will contribute a minimum of ten subjects per arm.
* Subjects will be assessed post-operatively during a minimum of five months after their second-eye surgery.
* Binocular defocus curves will be performed from +1.00 to -4.00 in 0.50 diopter steps and with +0.25 and -0.25 added.
* Self-reporting of visual complaints will be assessed.
* IOLSAT (IOL Satisfaction) and QUVID (Quality of Vision After Surgery) questionnaire will be administered at the study visit.
* Halo and Glare simulator VS Halo & Glare (visu-med.com) will be administered at the study visit.
* All visual acuity testing will be measured in LogMar and all study technicians and evaluators will be masked.
* PanOptix subjects will have been implanted with the toric and non-toric models.
* Synergy subjects will have been implanted with the toric and non-toric models.
* Demographic data will be collected to match the groups as closely as possible.

ELIGIBILITY:
Inclusion Criteria:

* Are willing and able to understand and sign an informed consent
* Are willing and able to complete all required study visits
* Are more than 40 years of age
* Patient diagnosed with cataracts both eyes and underwent uncomplicated cataract surgeries
* Patients with bilateral PanOptix (toric or non-toric)
* Patients with bilateral Synergy (toric or non-toric)
* Post-op best Corrected distance Visual Acuity for each eye is logMAR 0.1 (20/25) or better after cataract removal.
* Post-op residual refractive error +0.50 - -0.50 SE with ≤ 0.75 residual refractive astigmatism in each eye
* Minimum of two weeks post Yttrium Aluminum Garnet capsulotomy to treat posterior capsular opacification

Exclusion Criteria:

* Corneal dystrophies or degenerations
* Failure to return for follow up at designed intervals.
* Any conditions that might affect cataract removal (pseudoexfoliation, posterior polar cataract, Flomax, etc.)
* Any conditions during surgery that might prolong the cataract removal (capsular tear, inadequate pupil dilation, etc.)
* Strabismus with or without amblyopia in either eye
* Previous ocular surgery of any kind
* History of retinal detachment
* Any corneal abnormality, other than regular corneal astigmatism (as determined by corneal topography) that in the opinion of the investigator would confound the outcome(s) of the study
* Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that in the opinion of the investigator is clinically significant
* Subjects with glaucoma
* Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g. immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, etc)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with healthy eyes and uncomplicated bilateral implantation of Panoptix IOLs or Synergy IOLs.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Micheletti, MD, Principal Investigator — Berkeley Eye Center
Locations (1):
- Berkeley Eye Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Started | 153 | 77
Completed | 153 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy | Total
Number analyzed (Participants) | 153 | 77 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.3) | 65.9 (10.2) | 65.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 51 | 138
  Male | 66 | 26 | 92
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Binocular DCNVA (Distance Corrected Near Visual Acuity) at 40cm
Description: Binocular DCNVA Visual acuity testing will be measured in LogMar and all study technicians and evaluators will be masked. A summary of the data will be prepared for all subjects and categorized by the lens implanted. Variables measured on a continuous scale will be summarized to include sample size as well as the mean, standard deviation, median, minimum and maximum.
Time Frame: 3 months post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
logMAR | 0.03 (0.08) | 0.01 (0.07)

2. Secondary Outcome: Binocular Corrected Distance Visual Acuity (CDVA) Measured at 4m.
Description: Binocular CDVA measured at 4m. Visual acuity testing will be measured in LogMar and all study technicians and evaluators will be masked. A summary of the data will be prepared for all subjects and categorized by the lens implanted. Variables measured on a continuous scale will be summarized to include sample size as well as the mean, standard deviation, median, minimum and maximum.
Time Frame: 3 months post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
logMAR | -0.06 (0.06) | -0.07 (0.07)

3. Secondary Outcome: Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) Measured at 60cm.
Description: Binocular DCIVA measured at 60cm. Visual acuity testing will be measured in LogMar and all study technicians and evaluators will be masked. A summary of the data will be prepared for all subjects and categorized by the lens implanted. Variables measured on a continuous scale will be summarized to include sample size as well as the mean, standard deviation, median, minimum and maximum.
Time Frame: 3 months post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
logMAR | 0.00 (0.08) | 0.00 (0.07)

4. Secondary Outcome: Binocular Uncorrected Distance Visual Acuity (UDVA) Measured at 4m.
Description: Binocular UDVA measured at 4m. Visual acuity testing will be measured in LogMar and all study technicians and evaluators will be masked. A summary of the data will be prepared for all subjects and categorized by the lens implanted. Variables measured on a continuous scale will be summarized to include sample size as well as the mean, standard deviation, median, minimum and maximum.
Time Frame: 3 months post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
logMAR | -0.01 (0.08) | 0.00 (0.08)

5. Secondary Outcome: Binocular Uncorrected Intermediate Visual Acuity (UIVA) Measured at 60cm.
Description: Binocular UIVA measured at 60cm. Visual acuity testing will be measured in LogMar and all study technicians and evaluators will be masked. A summary of the data will be prepared for all subjects and categorized by the lens implanted. Variables measured on a continuous scale will be summarized to include sample size as well as the mean, standard deviation, median, minimum and maximum.
Time Frame: 3 months post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
logMAR | 0.00 (0.08) | 0.00 (0.08)

6. Secondary Outcome: Binocular Uncorrected Near Visual Acuity (UNVA) Measured at 40cm.
Description: Binocular UNVA measured at 40cm. Visual acuity testing will be measured in LogMar and all study technicians and evaluators will be masked. A summary of the data will be prepared for all subjects and categorized by the lens implanted. Variables measured on a continuous scale will be summarized to include sample size as well as the mean, standard deviation, median, minimum and maximum.
Time Frame: 3 months post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
logMAR | 0.03 (0.08) | 0.03 (0.08)

7. Secondary Outcome: Binocular Target Corrected Defocus Curve
Description: Binocular target corrected defocus curve. Visual acuity testing will be measured in LogMar and all study technicians and evaluators will be masked. A summary of the data will be prepared for all subjects and categorized by the lens implanted. Variables measured on a continuous scale will be summarized to include sample size as well as the mean, standard deviation, median, minimum and maximum.
Time Frame: 3 months post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
logMAR
  -3.00 D | 0.12 (0.09) | 0.09 (0.09)
  -2.50 D | 0.03 (0.08) | 0.03 (0.09)
  -2.00 D | -0.01 (0.08) | 0.01 (0.09)
  -1.50 D | 0.02 (0.09) | 0.02 (0.09)
  -1.00 D | 0.10 (0.09) | 0.06 (0.09)
  -0.50 D | 0.06 (0.07) | 0.03 (0.07)
  -0.25 D | -0.02 (0.07) | -0.04 (0.06)
  0.00 D | -0.07 (0.07) | -0.06 (0.06)
  0.25 D | -0.03 (0.07) | -0.01 (0.08)
  0.50 D | 0.04 (0.07) | 0.04 (0.09)
  1.00 D | 0.22 (0.10) | 0.21 (0.11)

8. Secondary Outcome: Patient Reported Satisfaction by IOLSAT Questionnaire.
Description: Patient reported satisfaction by IOLSAT questionnaire will be assessed. Variables measured on a categorical scale will be summarized to provide the number and percentage of subjects who provided each score. The percentage of patients "Satisfied" or "Very Satisfied" will be added for a total satisfaction percentage.
Time Frame: 3 months post operatively
Measure: Number; unit: percentage of participants
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
percentage of participants | 89 | 94

9. Secondary Outcome: Patient Reported Dysphotopsias Questionnaire (QUVID).
Description: Patient reported disphotopsias by QUVID questionnaire will be assessed. Variables measured on a categorical scale will be summarized to provide the number and percentage of subjects who provided each score. The percentage of subjects that answered "Never" for frequency are provided.
Time Frame: 3 months post operatively
Measure: Number; unit: percentage of participants
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
percentage of participants
  Starbursts | 65 | 49
  Halos | 38 | 38
  Glare | 48 | 55
  Haze | 84 | 86
  Blurred Vision | 87 | 75
  Double Vision | 97 | 100
  Dark Area | 98 | 96

10. Secondary Outcome: Post Operative Refraction, Manifest Refraction Spherical Equivalent (MRSE).
Description: Post operative refraction. A summary of the data will be prepared for all subjects and categorized by the lens implanted. Variables measured on a continuous scale will be summarized to include sample size as well as the mean, standard deviation, median, minimum and maximum.
Time Frame: 3 months post operatively
Measure: Mean (Standard Deviation); unit: D
Units Other Than Participants: eyes
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
Number analyzed (eyes) | 206 | 144
D | 0.24 (0.26) | 0.23 (0.26)

11. Other Pre Specified Outcome: Spectacle Independence Utilizing the IOLSAT.
Description: Spectacle independence utilizing the IOLSAT will be assessed. Variables measured on a categorical scale will be summarized to provide the number and percentage of subjects who provided each score. Spectacle independence was defined as answering "Never" or "Rarely" on the IOLSAT, the data presented is the percentage of subjects answering "Never" or "Rarely".
Time Frame: 3 months post operatively
Measure: Number; unit: percentage of participants
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
percentage of participants
  Overall | 92 | 97
  Distance | 99 | 100
  Intermediate | 99 | 100
  Near | 93 | 96

12. Other Pre Specified Outcome: Binocular Distacne Corrected Near Visual Acuity (DCNVA) at 33cm.
Description: Binocular DCNVA at 33cm. Visual acuity testing will be measured in LogMar and all study technicians and evaluators will be masked. A summary of the data will be prepared for all subjects and categorized by the lens implanted. Variables measured on a continuous scale will be summarized to include sample size as well as the mean, standard deviation, median, minimum and maximum.
Time Frame: 3 months post operatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
Number analyzed (Participants) | 153 | 77
logMAR | 0.09 (0.09) | 0.04 (0.08)

ADVERSE EVENTS:
Time Frame: 3 months postoperatively
Arm/Group | Alcon PanOptix | Johnson & Johnson Synergy
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/77
Other Adverse Events (participants affected / at risk) | 0/153 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT06041139/Prot_SAP_000.pdf